CLINICAL TRIAL: NCT02662010
Title: The Relationship of Advanced Glycation Endproducts in the Anterior Lens Capsule to Glycemic Status and Diabetic Retinopathy: A Cross Sectional Study of Patients With and Without Type 2 Diabetes Mellitus Undergoing Cataract Surgery
Brief Title: The Relationship Between Advanced Glycation Endproducts and Diabetes
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-2029; UL1TR001082 (NIH)
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Diabetic Retinopathy; Type 2 Diabetes Mellitus
Keywords: AGEs; glycemic control; T2DM
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Buffy Coat
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The overall purpose of this COMIRB application is to perform a cross-sectional pilot study to aid in the design of a prospective epidemiologic study for an NIH grant application. The long term goal of this research is to determine if AGEs are predictors of glycemic control and the development of diabetic retinopathy in patients with T2DM. Understanding these relationships could lead to a prospective prediction of the onset/worsening of diabetic retinopathy in T2DM patients and in pre-diabetic individuals.

DETAILED DESCRIPTION:
Below are the specific aims and research hypotheses for the pilot study:

Specific Aim 1: To successfully recruit 80 subjects (40 with no diabetes, 20 with diabetes and no diabetic retinopathy and 20 with diabetes and diabetic retinopathy) and obtain adequate samples (blood and lens capsule) for further testing.

Hypothesis 1:

Recruitment of subjects with and without diabetes and diabetic retinopathy is feasible within our clinic and the process for collecting, processing and storing samples is adequate to support the full study.

Specific Aim 2: To measure anterior lens capsule AGEs and HbA1c levels in recruited patients.

Hypothesis 2:

Levels of AGEs and HbA1c will be quantifiable in collected samples.

The pilot study aims are necessary to determine the feasibility of the full study, as well as to provide estimates of the (1) proportion of non-diabetic subjects with Abnormal HbA1c, (2) effect sizes and (3) variances for planning the full study.

The planned specific aims and research hypotheses for the full study are as follows:

Specific Aim 1: To determine whether anterior lens capsule AGEs differ in patients with and without a clinical diagnosis of T2DM.

Hypothesis 1:

Levels of AGEs will be higher in patients with a clinical diagnosis of T2DM compared with patients without a clinical diagnosis of diabetes.

Specific Aim 2: To determine if levels of AGEs measured from the anterior lens capsule are correlated with levels of Hemoglobin A1c (HbA1c) in patients without T2DM.

Hypothesis 2:

Levels of HbA1c will positively correlate with levels of HbA1c in all patients.

Specific Aim 3: To determine among patients with T2DM if levels of AGEs measured from the anterior lens capsule are higher in the group with diabetic retinopathy compared with the group with no diabetic retinopathy.

Hypothesis 3:

That among patients with T2DM: Levels of AGEs will be higher in the patients with diabetic retinopathy compared with the patients with no diabetic retinopathy.

AGEs are elevated in patients with diabetes (1, 3) and are reported to have a role in diabetic complications. (4, 5) Hyperglycemia results in higher intracellular glucose levels and the formation of metabolites from many complex interactions which in turn increase the production of AGEs. AGEs are a source of reactive oxygen species (ROS) with results in oxidative stress to tissues.(4) As reported, oxidative stress plays an important role in the microvascular and cardiovascular pathologic processed described in T2DM. (6) Importantly, oxidative stress is causal in the development of b cell dysfunction and insulin resistance, the two hallmarks of T2DM. (4)

ELIGIBILITY:
Inclusion criteria (cases):

* T2DM as documented by the referring physician, an HbA1C level of greater than 5.7 mmol/mol, or on T2DM medications beyond Metformin.
* 50% of the cases will have diabetic retinopathy as documented by the attending ophthalmologist and 50% will have no retinopathy.
* Age 60-80 years old.

Inclusion criteria (controls):

1. Normal HbA1C

   * No diabetes as documented by the referring physician, a HbA1C level of less than or equal to 5.7 mmol/mol, or not taking medications for T2DM with the exception of Metformin.
   * Age 60-80 years old.
2. Abnormal HbA1C

   * No diabetes as documented by the referring physician, a HbA1C level between 5.7 and 6.5 mmol/mol, and not taking medications for T2DM with the exception of Metformin.
   * Age 60-80 years old.

Exclusion criteria (cases):

* Type 1 diabetes as documented by the referring physician.
* <60 years old or >80 years old.
* If the patient has bilateral cataract surgery, the second surgery will be excluded
* Patients who have active cancer, being treated (receiving Chemotherapy or Radiation therapy) or disseminated, recent CVD event, MI or CVA within 6 months, and disease related weight loss of more than 10% in the past 3-6 months.

Exclusion criteria (controls):

* Type 1 or T2DM as documented by the referring physician.
* <60 years old or >80 years old.
* No treatment with Metformin or modifiers for risk of T1DM
* If the patient has bilateral cataract surgery, the second surgery will be excluded
* Patients who have active cancer, being treated (receiving Chemotherapy or Radiation therapy) or disseminated, recent CVD event, MI or CVA within 6 months, and disease related weight loss of more than 10% in the past 3-6 months.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Investigators propose recruiting 80 subjects (40 with no diabetes, 20 with diabetes and no diabetic retinopathy and 20 with diabetes and diabetic retinopathy).
  Within the 40 control patients without a clinical diagnosis of T2DM, 20 will have an abnormal HbA1C at the time of surgery. It is important to enroll the patients with an abnormal HbA1C in order to see if there are early manifestations of an abnormal glucose level as detected by AGEs in the anterior lens capsule.
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Change in Advanced Glycation Endproducts (AGE) Levels | 1 year

SECONDARY OUTCOMES:
Change in HbA1C Levels | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ram Nagaraj, PhD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- Universtiy of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milne R, Brownstein S. Advanced glycation end products and diabetic retinopathy. Amino Acids. 2013 Jun;44(6):1397-407. doi: 10.1007/s00726-011-1071-3. Epub 2011 Sep 11. PMID 21909978
- [Background] Ulrich P, Cerami A. Protein glycation, diabetes, and aging. Recent Prog Horm Res. 2001;56:1-21. doi: 10.1210/rp.56.1.1. PMID 11237208
- [Background] Yan SF, D'Agati V, Schmidt AM, Ramasamy R. Receptor for Advanced Glycation Endproducts (RAGE): a formidable force in the pathogenesis of the cardiovascular complications of diabetes & aging. Curr Mol Med. 2007 Dec;7(8):699-710. PMID 18331228
- [Background] Nowotny K, Jung T, Hohn A, Weber D, Grune T. Advanced glycation end products and oxidative stress in type 2 diabetes mellitus. Biomolecules. 2015 Mar 16;5(1):194-222. doi: 10.3390/biom5010194. PMID 25786107
- [Background] Monnier VM, Sell DR, Genuth S. Glycation products as markers and predictors of the progression of diabetic complications. Ann N Y Acad Sci. 2005 Jun;1043:567-81. doi: 10.1196/annals.1333.065. PMID 16037280
- [Background] Giacco F, Brownlee M. Oxidative stress and diabetic complications. Circ Res. 2010 Oct 29;107(9):1058-70. doi: 10.1161/CIRCRESAHA.110.223545. PMID 21030723
- [Background] Smuda M, Henning C, Raghavan CT, Johar K, Vasavada AR, Nagaraj RH, Glomb MA. Comprehensive analysis of maillard protein modifications in human lenses: effect of age and cataract. Biochemistry. 2015 Apr 21;54(15):2500-7. doi: 10.1021/bi5013194. Epub 2015 Apr 7. PMID 25849437